CLINICAL TRIAL: NCT02224989
Title: A Pilot Feasibility Study of a Novel Mind-body Intervention Program for Veterans With PTSD
Brief Title: Mind-Body Intervention for Veterans With PTSD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: 1) Difficulties in recruiting veterans and 2) the funding was used up completely
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Yoshio Nakamura, Research Associate Professor, University of Utah
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB_00052611
Record Dates: First submitted 2014-08-21; First posted 2014-08-25 (Estimated); Last update posted 2018-05-07 (Actual); Status verified 2018-05

CONDITIONS: Stress Disorders, Post-Traumatic
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mind-Body Bridging (Experimental): An awareness training program using mindfulness-based techniques.
  Interventions: Behavioral: Mind-Body Bridging

INTERVENTIONS:
Behavioral: Mind-Body Bridging — An awareness training program. One 2 hr class per week for 10 weeks.

SUMMARY:
This pilot project evaluates the efficacy of a mind-body awareness training intervention, Mind-Body Bridging (MBB), in veteran patients with PTSD and comorbid symptoms. Evidence for relative therapeutic benefit will be indicated by the difference in outcomes from pre- to post-intervention for PTSD as the primary outcome.

DETAILED DESCRIPTION:
PTSD is a difficult illness to treat and there is a lack of interventions that effectively reduce it. In recent years, attention has focused on treating PTSD patients by including a sleep-focused intervention since those with PTSD, such as military personnel, almost always report some form of sleep disturbance (Neylan et al. 1998; Lewis et al. 2009). In fact, since sleep disturbance is so prevalent in PTSD, it is considered a hallmark of PTSD diagnosis (Ross et al. 1989). Two classical PTSD symptoms, hyperarousal and re-experiencing the traumatic event, comprise sleep difficulty and nightmares, respectively (Lamarche and De Koninck 2007). Preliminary evidence suggests that interventions targeting sleep may be beneficial in the treatment of PTSD (Germain et al. 2007; Swanson et al. 2009; Nakamura et al. 2011).

This study will evaluate the effectiveness of mind-body bridging (MBB) as a primary group psychotherapy treatment for reduction of PTSD symptoms among veterans. MBB is an awareness training program,(Block and Block 2007) which has been recently developed into a workbook specifically for PTSD (Block and Block 2010). MBB has been used successfully at the George E. Wahlen Veterans Affairs Medical Center (VAMC) for more than 5 years as an adjunctive treatment. MBB is well accepted by veterans and anecdotally has been reported to improve mood as well as PTSD and other anxiety symptoms. Furthermore, published pilot studies have provided preliminary evidence of its benefits.(Tollefson et al. 2009; Nakamura et al. 2011). In particular, Nakamura et al.(2011) tested a brief sleep-focused MBB intervention program in a randomized controlled trial, which demonstrated improved sleep and decreased PTSD symptoms. Our clinical experience and these preliminary studies indicate that a pilot feasibility study of MBB as a specific treatment for PTSD is warranted.

The proposed, non-randomized single-group study of MBB will serve as a pilot feasibility study investigating a 10-week MBB program offered to veterans who are clinically diagnosed to suffer from PTSD. In this pilot study, we determine whether MBB is a beneficial intervention program for PTSD and co-morbidities, including insomnia, depression, etc., based on self-report measures and clinical evaluations.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion of subjects will be based on: pre-screening score of 50 or greater on the PTSD Checklist for Military (PCL-M). Since we are also interested in the effects of MBB on co-morbid illnesses besides PTSD, we will include subjects who present with other behavioral health conditions, including sleep disturbance, depression, anxiety, pain, and any general medical conditions, except as defined as exclusion criteria. Subjects using anti-anxiety, anti-depressants, sleep and pain medications, and other medications for any condition that is not under exclusion criteria will be admitted to the study. Participants must be willing to commit to the 10-week course and complete all outcome measures, be literate in English and able to provide informed consent.

Participants will be asked to refrain from engaging in other PTSD treatment programs for the duration of the proposed study, but can remain on their medications and continue with their usual medical or mental health care. They will also be allowed to continue with other activities (such as physical exercise, meditation, yoga, etc.), which they may have already incorporated into their life.

Exclusion Criteria:

* A patient will be excluded from the study under the following conditions:

  1. currently enrolled in active PTSD treatment program.
  2. identifying with major psychopathology (i.e., schizophrenia, mania, or poorly controlled bipolar disorder, borderline or antisocial personality disorder) and was psychiatrically hospitalized within the past 90 days.
  3. cognitive impairment or dementia.
  4. severe medical disease such as uncontrolled hypertension or diabetes, or terminal illness, e.g., cancer.
  5. active substance abuse disorder
  6. suicidal ideation with intent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Change in the self-report measure of PTSD using the PTSD Checklist for Military (PCLM), from baseline to 3 month follow-up. | Baseline, 5 weeks (mid-treatment), 10 weeks (post-treatment), 3 month follow-up
  The PCL-M is a well-validated 17-item self-report measure to assess PTSD severity among military personnel; both male and female, to assess military-related PTSD. Reliability evidence is very good. Items are based on the Diagnostic and Statistical Manual-IV (DSM-IV) criteria, and are rated on a 5-point Likert-type scale that allows the derivation of a quantifiable total score.

SECONDARY OUTCOMES:
Change in subjective measure of sleep using the Medical Outcomes Study - Sleep Scale (MOS-SS), from baseline to 3-month follow-up. | Baseline, 5 weeks (mid-treatment), 10 weeks (post-treatment), 3-month follow-up
  The MOS-SS is a 12-item validated questionnaire evaluating sleep outcomes over the past 7 days. The MOS-SS provides an index of sleep problems, including sleep disturbance, sleep adequacy, daytime somnolence, snoring, waking up short of breath with a headache, and quantity of sleep. The MOS-SS was validated as a retrospective assessment of sleep performance over the previous 4 weeks, and compares favorably with the Pittsburgh Sleep Quality Index (PSQI). We have used a modified version of MOS-SS to assess the subject's sleep patterns over the previous 7 days.
Change in subjective measure of resilience using the Response to Stressful Experience Scale (RSES), from baseline to 3-month follow-up. | Baseline, 5 weeks (mid-treatment), 10 weeks (post-treatment), 3-month follow-up
  The RSES is a multidimensional measure of resilience validated in a large sample of active-duty and reserve military personnel. This 22-item scale demonstrates good internal consistency. Confirmatory factor analysis revealed reasonable fit for a model of resilience comprising six-dimensions: (1) Cognitive Flexibility, (2) Spirituality, (3) Active Coping, (4) Self-efficacy, (5) Making-meaning, and (6) Restoration. The major strength of this scale is that it is indexed to a specific traumatic or extremely stressful event, such as combat and operational stress in military personnel. .
Change in subjective measure of Health Related Quality of Life using the Medical Outcomes Study SF-36 for Veterans (VR-36), from baseline to 3-month follow-up. | Baseline, 5 weeks (mid-treatment), 10 weeks (post-treatment), 3-month follow-up
  Medical Outcomes Study Short Form-36 (SF-36) for Veterans (VR-36). The VR-36 is a modification of the original SF-36, adapted for Veterans. It consists of the same eight sections as the SF-36. The instrument provides a global score, as well as the following subscale scores: functional capacity, physical aspects, pain, general health condition, vitality, social aspects and emotional aspects, and mental health.
Change in subjective measure of depression using the Center for Epidemiologic Studies Depression Scale (CES-D), from baseline to 3-month follow-up. | Baseline, 5 weeks (mid-treatment), 10 weeks (post-treatment), 3-month follow-up
  The CES-D is one of the most common validated screening tests for helping an individual to determine his or her depression quotient. The 20-item test measures depressive feelings and behaviors during the past week.
Change in subjective measure of mindfulness using the Five-facet Mindfulness Questionnaire (FFMQ), from baseline to 3-month follow-up. | Baseline, 5 weeks (mid-treatment), 10 weeks (post-treatment), 3-month follow-up
  The FFMQ includes 39 items and assesses five distinct, interpretable facets of mindfulness, including: 1) observing, 2) describing, 3) acting with awareness, 4) non-judging of inner experience, and 5) non-reactivity to inner experience.
Change in subjective measure of well-being using the Well-Being Index (WBI), from baseline to 3-month follow-up. | Baseline, 5 weeks (mid-treatment), 10 weeks (post-treatment), 3-month follow-up
  The WBI is a five item scale evaluating both positive and negative aspects of emotional functioning, developed and validated by the World Health Organization Collaborating Centre in Mental Health.
Change in subjective measure of health-related quality of life using the Medical Outcomes Study Short Form - 12 (SF-12), from baseline to 3-month follow-up. | Baseline, 5 weeks (mid-treatment), 10 weeks (post-treatment), 3-month follow-up
  The SF-12 is a much shortened version of the SF-36, comprising 12 items. It will be measured on a weekly basis.
Change in subjective measure of quality of life using the Mind-Body Bridging Quality of Life scale (MBB QOL), from baseline to 3-month follow-up. | Baseline, 5 weeks (mid-treatment), 10 weeks (post-treatment), 3-month follow-up
  The MBB QOL is a non-validated questionnaire used to assess the effects of MBB on quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Yoshio Nakamura, Ph.D., Principal Investigator — University of Utah
Locations (1):
- Salt Lake City Veterans Affairs Health Care System, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No